CLINICAL TRIAL: NCT05199948
Title: Weight, Energy, Lipids, and the Liver (WELL) Study: Dietary Fat Quality and Ectopic Lipids in the Liver
Brief Title: Weight, Energy, Lipids, and the Liver (WELL) Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Martha Belury, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021H0290
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soybean Oil (Experimental): Consumption of study foods each day made with soybean oil
  Interventions: Other: Soybean Oil Foods
- Palm Oil (Placebo Comparator): Consumption of study foods each day made with palm oil
  Interventions: Other: Palm Oil Foods

INTERVENTIONS:
Other: Soybean Oil Foods — Three food product containing 10g of soybean oil each will be consumed each day for a today of 30g of soybean oil consumed each day
  Arms: Soybean Oil
Other: Palm Oil Foods — Three food product containing 10g of palm oil each will be consumed each day for a today of 30g of palm oil consumed each day
  Arms: Palm Oil

SUMMARY:
The research study is a parallel arm, randomized placebo-controlled clinical trial designed to assess changes in hepatic lipid accumulation, visceral adipose tissue and postprandial lipid, markers of inflammation and energy metabolism in participants who consume 3 study foods per day for 16 week, while maintaining their body weight.

DETAILED DESCRIPTION:
The study objectives include:

1. To determine the impact of dietary soybean oil on ectopic liver fat and visceral adipose in adults with nonalcoholic fatty liver disease (NAFLD) or similar diagnosis
2. To evaluate the effect of soybean oil supplementation on postprandial lipids, markers of inflammation and energy metabolism
3. To measure the strength of the association of change in plasma linoleic acid with changes in ectopic liver fat, visceral adipose, and postprandial lipids, markers of inflammation and energy metabolism
4. To explore emerging mechanistic targets of LA-rich soybean oils that are linked with reduced liver fat and better cardiometabolic health

ELIGIBILITY:
Inclusion Criteria:

* Nonalcoholic fatty liver disease (NAFLD), Nonalcoholic Steatohepatitis (NASH) or similar
* Body Mass Index of 20-55 kg/m2

Exclusion Criteria:

* Unstable management of heart failure, heart disease events within 3 months, a need for heart surgeries or procedures, and/or the use of a pacemaker or defibrillator
* Current or previous diagnosis of severe kidney failure or diseases, some liver and pulmonary diseases
* Severe or uncontrolled circulatory diseases and autoimmune diseases
* Current diagnosis of or current treatment of cancer other than non-melanoma skin cancer
* Current or previous diagnosis of type 1 diabetes
* Use of Vitamin E supplements or Actos and Glucagon-like Peptide-1 medications for less than 1 months prior to enrolling.
* Gastrointestinal diseases or disorders (including pancreatic and gastric bypass surgery) that would prevent participants from tolerating the study foods
* Food Allergy or intolerances
* Any dietary restriction where consumption of the study foods, study meals/snack or meal challenge or any ingredient would be contraindicated
* Use of medications where consuming the food products would be contraindicated
* Use of supplements high in linoleic acid in the past 4 weeks prior to enrolling
* Hyperthyroidism
* Pregnancy and lactation
* Alcohol or drug abuse
* Inability to access veins for venipuncture
* Claustrophobia
* Metal implants or metallic foreign objects in the body

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in ectopic liver lipids | Week 0 and Week 16
  To determine the impact of dietary soybean oil on ectopic liver fat measured through MRI

SECONDARY OUTCOMES:
Changes in visceral adipose tissue | Week 0 and Week 16
  To determine the impact of dietary soybean oil on visceral adipose tissue measured through MRI
Changes in postprandial lipids | Week 0 and Week 16
  To evaluate the effect of soybean oil supplementation on postprandial lipid panel including total cholesterol, HDL-Cholesterol, LDL-Cholesterol, Triglycerides
Changes in postprandial markers of inflammation | Week 0 and Week 16
  To evaluate the effect of soybean oil supplementation on the postprandial IL-6, Tumor necrosis factor, and C-reactive protein in the blood
Changes in postprandial energy metabolism | Week 0 and Week 16
  To evaluate the effect of soybean oil supplementation on postprandial indirect calorimetry or respiratory gas exchange

OTHER OUTCOMES:
Association of changes in plasma linoleic acid with ectopic liver lipids, visceral adipose tissue, and postprandial lipids, markers of inflammation and energy metabolism | Week 0 and Week 16
  Use multiple linear regressions to determine the association of change in plasma linoleic acid with changes in ectopic liver fat, visceral adipose, and postprandial total cholesterol, HDL-Cholesterol, LDL-Cholesterol, Triglycerides, L-6, Tumor necrosis factor, and C-reactive protein and indirect calorimetry
Changes in cardiolipin species | Week 0 and Week 16
  To determine the impact of dietary soybean oil on peripheral blood mononuclear cell cardiolipin species measured using electrospray ionization-mass spectrometry coupled to high-performance liquid chromatography
Changes in mitochondria function | Week 0 and Week 16
  To determine the impact of dietary soybean oil on peripheral blood mononuclear cell mitochondria oxygen consumption rate using the seahorse assay

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Human Nutrition Laboratory, Columbus, Ohio, United States